CLINICAL TRIAL: NCT01809652
Title: Remote Implant Support
Brief Title: Feasibility Study of Remote Support for Implantable Pulse Generator (IPG)/Implantable Cardioverter Defibrillator (ICD) Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Remote Implant Support
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Bradycardia; Sudden Cardiac Arrest
Keywords: Pacemaker; Defibrillator; Remote Consultation
MeSH Terms: conditions — Bradycardia; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remote Implant Support (Experimental): Implant supported through remote implant support capability
  Interventions: Other: Remote Implant Support Capability

INTERVENTIONS:
Other: Remote Implant Support Capability — Use of audio and video telepresence and remote control of device programmer to allow implant to be supported from a remote location

SUMMARY:
The purpose of this study is to gain real world, live implant experience with the remote implant support system. This system is intended to provide the technical support for device implants from a remote location through telepresence (audio and video) and remote control. Specifically, the goals of this study are to corroborate bench testing, assess the performance of the system, gain understanding of the workflows, customer experience, and logistics.

The intent of the remote support model is to provide the same support that would typically be provided by a local support person, only remotely. As such, the remote support person would only perform actions that a local support person would routinely do under the direction of a physician. This may involve observing patient data, providing technical support and advice, and performing testing and device reprogramming via remote control of the programmer.

ELIGIBILITY:
Inclusion Criteria:

* Planned IPG implant or planned ICD (without CRT) implant
* Signed informed consent

Exclusion Criteria:

* Pacing dependency
* Defibrillation threshold testing planned
* Basal ventricular rate >110 beats per minute
* Younger than 18 years
* Pregnant
* Currently involved in another IPG or ICD related clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
System Integrity | At implant
  Percentage of patients whose implantable devices with clinically equivalent programming by remote support and local support.
Successful Support | At implant
  Percentage of implant attempts with successful support. If the local support person does not participate in any part of the surgery, other than observing, then the remote support will be called a success.

CONTACTS AND LOCATIONS:
Locations (1):
- Centennial Heart, Nashville, Tennessee, United States